CLINICAL TRIAL: NCT07237542
Title: Effect of Remote Ischemic Preconditioning on Early Neurological Deterioration in Acute Perforating Artery Infarction (RIC-END): A Randomised Multicentre Trial
Brief Title: Effect of Remote Ischemic Preconditioning on Early Neurological Deterioration in Acute Perforating Artery Infarction
Acronym: RIC-END
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Xinfeng Liu, Professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIC-END
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke; Remote Ischaemic Preconditioning
Keywords: perforating artery stroke; remote ischemic preconditioning; early neurological deterioration; randomized controlled trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Masking Description: open label, blinded outcome assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): The standard RIC procedure involves placing a blood pressure cuff on both upper limbs, rapidly inflating the cuff to occlude arterial blood flow and induce transient limb ischemia, followed by deflating the cuff to restore blood perfusion. RIC is administered twice daily on both upper limbs, with each session consisting of 5 cycles, for 5-7 consecutive days. The inflation pressure for RIC treatment is set at 200 mmHg.
  Interventions: Device: remote ischemic preconditioning
- shame RIC group (Sham Comparator): The standard RIC procedure involves placing a blood pressure cuff on both upper limbs, rapidly inflating the cuff to occlude arterial blood flow and induce transient limb ischemia, followed by deflating the cuff to restore blood perfusion. RIC is administered twice daily on both upper limbs, with each session consisting of 5 cycles, for 5-7 consecutive days. The inflation pressure for RIC treatment is set at 60 mmHg.
  Interventions: Device: sham remote ischemic preconditioning

INTERVENTIONS:
Device: remote ischemic preconditioning — The standard RIC procedure involves placing a blood pressure cuff on both upper limbs, rapidly inflating the cuff to occlude arterial blood flow and induce transient limb ischemia, followed by deflating the cuff to restore blood perfusion. RIC is administered twice daily on both upper limbs, with each session consisting of 5 cycles, for 5-7 consecutive days. The inflation pressure for RIC treatment is set at 200 mmHg.
  Arms: RIC group
Device: sham remote ischemic preconditioning — The standard RIC procedure involves placing a blood pressure cuff on both upper limbs, rapidly inflating the cuff to occlude arterial blood flow and induce transient limb ischemia, followed by deflating the cuff to restore blood perfusion. RIC is administered twice daily on both upper limbs, with each session consisting of 5 cycles, for 5-7 consecutive days. The inflation pressure for RIC treatment is set at 60 mmHg.
  Arms: shame RIC group

SUMMARY:
This study aims to conduct a prospective, randomized, double-blind, multicenter, parallel-controlled, group-sequential trialto scientifically evaluate the safety and efficacy of remote ischemic preconditioning (RIC) in preventing early neurological deterioration (END) in patients with acute perforating artery infarction (PAI).

DETAILED DESCRIPTION:
Penetrating artery infarction (PAI) is a single small deep infarct within the territory of a perforating artery, accounting for 15.3%-25% of all ischemic strokes. Early neurological deterioration (END) is a critical factor contributing to poor prognosis in PAI. END is generally defined as an increase of ≥2 points on the National Institutes of Health Stroke Scale (NIHSS) within 7 days after stroke onset. Remote ischemic preconditioning (RIC) involves repeated, low-intensity ischemic training of both upper limbs to enhance the resistance of organs to severe ischemic injury. RIC confers protective effects on ischemic brain tissue and may serve as a new therapeutic approach for intracranial atherosclerosis and acute cerebral infarction. However, large-scale randomized controlled trials evaluating the clinical efficacy of RIC in acute PAI are lacking. Therefore, this study aims to conduct a multicenter, prospective, randomized clinical trial to scientifically assess the clinical efficacy of RIC in patients with acute PAI, providing evidence-based support for its application in this population.

In this trial, patients with acute PAI (within 48 hours from onset to randomization) will be included. In the screening stage, participants who meet the trial's inclusion criteria-after completing screening/baseline assessment and signing the informed consent-will be randomly assigned in a 1:1 ratio to one of the following two treatment groups: the experimental group will receive RIC (200 mmHg), and the control group will receive sham RIC (60 mmHg). The primary end point is the incidence of END within 5 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Diagnosed with acute ischemic stroke;
3. Clinical symptoms consistent with perforating artery infarction (NIHSS score ≤5, with consciousness item 1a ≤1);
4. Time from onset to randomization within 48 hours;
5. Diffusion-weighted imaging (DWI) showing a single infarct in the perforating artery territory with a maximum diameter ≤30 mm, meeting at least one of the following:

(1) Diameter ≤15 mm and involving two or more axial slices; (2) Maximum diameter ≥15 mm; (3) Connected to the ventral surface of the pons but not crossing the midline; 6) Stenosis of parent artery <70%; 7) Signed informed consent obtained from the patient or their legally authorized representative.

Exclusion Criteria:

1. Received intravenous thrombolysis or endovascular treatment prior to randomization;
2. Secondary stroke caused by brain tumor, traumatic brain injury, hematologic disorders, or other conditions;
3. History of intracranial hemorrhage;
4. Presence of RIC contraindications, such as severe upper limb soft tissue injury, fracture, subclavian artery stenosis, or peripheral vascular disease;
5. Uncontrolled severe hypertension (systolic blood pressure [BP] ≥180 mmHg or diastolic BP ≥110 mmHg);
6. Severe hepatic or renal dysfunction (Alanine Aminotransferase or Aspartate Aminotransferase > 3 × upper limit of normal; creatine kinase >3 × upper limit of normal; estimated Glomerular Filtration Rate < 30 mL / min / 1.73 m²);
7. Patients with thrombocytopenic purpura, coagulation disorders, or active visceral bleeding;
8. Patients in the acute phase of fundus hemorrhage;
9. History of severe aphasia or psychiatric disorders affecting clinical assessment;
10. Life expectancy <90 days;
11. Pregnancy;
12. Inability to comply with follow-up;
13. Participation in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 910 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of early neurological deterioration | 5 days after randomization
  an increase of ≥2 points in the National Institutes of Health Stroke Scale (NIHSS), including an increase of ≥1 point in the motor score. NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits).

SECONDARY OUTCOMES:
The incidence of early neurological deterioration | 2 days after randomization
  an increase of ≥2 points in the National Institutes of Health Stroke Scale (NIHSS), including an increase of ≥1 point in the motor score. NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits).
Proportion of patients with a modified Rankin Scale score of 0-1 | 90 days after randomization
  modified Ranking score: ranging from 0 to 6, with higher values indicating a worse functional outcome.
The incidence of early neurological improvement | 5 days after randomization
  defined as a decrease of ≥2 points in National Institutes of Health Stroke Scale (NIHSSS). NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits).
The incidence of early neurological improvement | 2 days after randomization
  defined as a decrease of ≥2 points in National Institutes of Health Stroke Scale (NIHSS). NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits).
The incidence of major adverse cardiovascular events | 90 days after randomization
  Major adverse cardiovascular events (MACE) refers to a composite measure of serious cardiovascular complications, typically including cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke, sometimes also encompassing hospitalization for unstable angina or urgent revascularization.
Barthel Index | 90 days after randomization
  Barthel Index is an ordinal disability score of 10 categories (range from 0 to 100, higher values indicate better prognosis)
EuroQol 5-Dimension 5-Level Questionnaire score | 90 days after randomization
  The EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L score) is a standardized index measuring a person's overall health-related quality of life, based on five dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-each rated on five levels of severity. EQ-5D-5L scores range from -0.59 to 1, where 1 is the best possible health state.

OTHER OUTCOMES:
The incidence of adverse events related to RIC | within 90 days from randomization
  Clinical safety endpoint
The incidence of mortality | within 90 days from randomization
  Clinical safety endpoint
The incidence of adverse events | within 90 days from randomization
  Clinical safety endpoint
The incidence of severe adverse events | within 90 days from randomization
  Clinical safety endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Medical School of Nanjing University, Nanjing, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No